CLINICAL TRIAL: NCT03543371
Title: Neuropsychological Outcome After Cardiac Arrest: A Prospective Case Control Sub-study of the Targeted Hypothermia Versus Targeted Normothermia After out-of Hospital Cardiac Arrest Trial (TTM2)
Brief Title: Neuropsychological Outcome After Cardiac Arrest
Status: Completed | Type: Observational
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other); Halmstad County Hospital (Other); Sahlgrenska University Hospital (Other); Mid and South Essex NHS Foundation Trust (Other); Cardiff and Vale University Health Board (Other Government); Aarhus University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CardiacArrestLundNeuropsych
Record Dates: First submitted 2018-05-17; First posted 2018-06-01 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2023-09

CONDITIONS: Heart Arrest, Out-Of-Hospital; Hypoxia-Ischemia, Brain; Cognition Disorders; Psychological Distress; Fatigue; Insomnia
Keywords: Neuropsychology
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Hypoxia-Ischemia, Brain; Cognition Disorders; Fatigue; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cardiac Arrest survivors: Cardiac arrest survivors at selected TTM2-sites only.
  Interventions: Diagnostic Test: Neuropsychological assessment
- Myocardial Infarction patients: A control group from a cohort of patients with myocardial infarction with performed coronary angiography but no occurrence of cardiac arrest will be recruited at 1:1 ratio.
  Interventions: Diagnostic Test: Neuropsychological assessment

INTERVENTIONS:
Diagnostic Test: Neuropsychological assessment — Standardized neuropsychological battery consisting of the following tests and questionnaires: Wechsler Adult Intelligence Scale - Fourth Edition (WAIS-IV) Vocabulary, Delis-Kaplan Executive Function System (D-KEFS) Verbal Fluency, WAIS-IV Block Design, WAIS-IV Matrix Reasoning, WAIS-IV Digit Span, Wechsler Memory Scale - Third Edition (WMS-III) Spatial Span, Rey Auditory Verbal Learning Test (RAVLT), WMS-III Logical Memory, Brief Visuospatial Memory Test-Revised (BVMT-R), Trail Making Test (TMT) A & B, D-KEFS Color Word Interference Test, Behavioral Assessment of the Dysexecutive Syndrome Dysexecutive Questionnaire (BADS DEX), Multidimensional Fatigue Inventory (MFI-20), Minimal Insomnia Symptom Scale (MISS), Hospital Anxiety and Depression Scale (HADS).

SUMMARY:
This study is a sub-study to the large pragmatic Target Temperature Management 2 Trial (TTM2-trial, ClinicalTrials.gov Identifier: NCT02908308), assessing effectiveness of controlled hypothermia after out-of-hospital cardiac arrest (OHCA).

This study is designed to provide detailed information on cognition after OHCA and its relationship to associated factors as emotional function, fatigue, and sleep. A secondary aim is to utilize this information to validate a neurocognitive screening battery used 6 months after OHCA in the TTM2-trial.

Approximately 7 and 24 months after OHCA, survivors at selected TTM2 study sites will perform a standardized neuropsychological assessment including performance-based tests of cognition and questionnaires of behavioral and emotional function, fatigue, and insomnia. At 1:1 ratio, a control group of myocardial infarction (MI) patients but no occurrence of cardiac arrest will be recruited and perform the same test battery. Group differences at 7 and 24 months will be analyzed per cognitive domain (verbal, visual/constructive, short-term working memory, episodic memory, processing speed, executive functions). Results of the OHCA survivors on the TTM2 neurocognitive screening battery will be compared with neuropsychological test results at 7 months time.

ELIGIBILITY:
Inclusion Criteria:

* OHCA of a presumed cardiac or unknown cause (OHCA cohort only)
* Sustained return of spontaneous circulation (ROSC) during intensive care - defined as 20 minutes with signs of circulation without the need for chest compressions (OHCA cohort only)
* Unconsciousness - defined as not being able to obey verbal commands (FOUR-score motor response of <4) and no verbal response to pain after sustained ROSC (OHCA cohort only)
* Inclusion within 180 minutes of ROSC (OHCA cohort only)
* During intensive care - eligible for intensive care without restrictions or limitations (OHCA cohort only)
* MI with performed coronary angiography (MI cohort only)

Exclusion Criteria:

* Temperature on admission <30°C (OHCA cohort only)
* On extracorporeal membrane oxygenation (ECMO) prior to return of spontaneous circulation (OHCA cohort only)
* Obvious or suspected pregnancy
* Intracranial bleeding (OHCA cohort only)
* Severe chronic obstructive pulmonary disorder (COPD) with long-term home oxygen therapy
* Clinical dementia diagnosis before the event
* Inability to speak the local language well enough to complete the assessment without assistance from an interpreter
* Inability to meet for a face-to-face examination
* Clinical Frailty Scale Index ≥8, indicating very severe frailty
* Cardiac arrest before or in connection with MI (MI cohort only)
* Active substance abuse

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: OHCA survivors at TTM2-sites participating in this study. Survivors are invited to partake in this study at the regular six-month follow-up of the TTM2-trial.
  The cohort of MI patients acting as controls are recruited and assessed at one participating site per country through quality registers.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2018-07-13 (Actual); Primary Completion 2021-01-11 (Actual); Study Completion 2022-05-23 (Actual)

PRIMARY OUTCOMES:
Cognitive impairment | 7 months after the cardiac event
  Cognitive function in OHCA and MI patients, using composite z-scores from the neuropsychological tests grouped by cognitive domain.

SECONDARY OUTCOMES:
Sensitivity and specificity of the neurocognitive screening battery in the main TTM2-trial | 7 months post-arrest
  Validation of the neurocognitive screening battery in OHCA patients, using the detailed neuropsychological test battery as a gold standard with sensitivity and specificity analyses. Here, patients will be considered to have a cognitive impairment if they meet any of the following criteria on the neuropsychological tests: 1) an impaired composite z-score defined as z ≤ - 1.65 in at least one cognitive domain; 2) z ≤ - 1.65 in at least two scores used for cognitive domain calculation. Cut-scores for indicated impairment on the neurocognitive screening battery will be < 26 on the MoCA, z≤-1 on the SDMT, ≥3.08 on the IQCODE-CA and the answer "no" to question 2 at the TSQ.

OTHER OUTCOMES:
Change in cognitive function | 7 months, 24 months after the cardiac event
  Longitudinal change in cognitive function in OHCA and MI patients, analyzed with a mixed model regression.

CONTACTS AND LOCATIONS:
Overall Officials: Niklas Nielsen, MD, PhD, Study Director — Lund University; Gisela Lilja, PhD, OT, Study Director — Lund University; Tobias Cronberg, MD, PhD, Study Director — Lund University; Susanna Vestberg, PhD, Lic.Psych., Study Director — Lund University; Erik Blennow Nordström, PhD, Lic.Psych., Principal Investigator — Lund University
Locations (8):
- Aarhus University Hospital, Aarhus, Denmark
- Sweden (5):
  - Sahlgrenska University Hospital, Gothenburg
  - Halmstad County Hospital, Halmstad
  - Helsingborg Hospital, Helsingborg
  - Skane University Hospital, Lund
  - Skane University Hospital, Malmo
- United Kingdom (2):
  - The Essex Cardiothoracic Centre, Basildon and Thurrock University Hospitals NHS Foundation Trust, Basildon, Essex
  - University Hospital of Wales, Cardiff and Vale University Health Board, Cardiff, Wales

REFERENCES:
- [Background] Blennow Nordstrom E, Lilja G, Vestberg S, Ullen S, Friberg H, Nielsen N, Heimburg K, Evald L, Mion M, Segerstrom M, Grejs AM, Keeble T, Kirkegaard H, Ljung H, Rose S, Wise MP, Rylander C, Unden J, Cronberg T. Neuropsychological outcome after cardiac arrest: a prospective case control sub-study of the Targeted hypothermia versus targeted normothermia after out-of-hospital cardiac arrest trial (TTM2). BMC Cardiovasc Disord. 2020 Oct 7;20(1):439. doi: 10.1186/s12872-020-01721-9. PMID 33028221
- [Result] Blennow Nordstrom E, Evald L, Mion M, Segerstrom M, Vestberg S, Ullen S, Heimburg K, Gregersen Oestergaard L, Grejs AM, Keeble TR, Kirkegaard H, Rylander C, Wise MP, Lilja G. Combined use of the Montreal Cognitive Assessment and Symbol Digit Modalities Test improves neurocognitive screening accuracy after cardiac arrest: A validation sub-study of the TTM2 trial. Resuscitation. 2024 Sep;202:110361. doi: 10.1016/j.resuscitation.2024.110361. Epub 2024 Aug 13. PMID 39147306
- [Result] Vig A, Vestberg S, Evald L, Mion M, Segerstrom M, Ullen S, Arestedt K, Nielsen N, Cronberg T, Lilja G, Blennow Nordstrom E. Psychometric properties of the Dysexecutive Questionnaire (DEX) in individuals with a previous cardiac event. Neuropsychol Rehabil. 2025 Nov 27:1-21. doi: 10.1080/09602011.2025.2591784. Online ahead of print. PMID 41308659
- [Result] Blennow Nordstrom E, Vestberg S, Evald L, Mion M, Segerstrom M, Ullen S, Bro-Jeppesen J, Friberg H, Heimburg K, Grejs AM, Keeble TR, Kirkegaard H, Ljung H, Rose S, Wise MP, Rylander C, Unden J, Nielsen N, Cronberg T, Lilja G. Neuropsychological outcome after cardiac arrest: results from a sub-study of the targeted hypothermia versus targeted normothermia after out-of-hospital cardiac arrest (TTM2) trial. Crit Care. 2023 Aug 26;27(1):328. doi: 10.1186/s13054-023-04617-0. PMID 37633944